CLINICAL TRIAL: NCT07218614
Title: Can Mobilizations Applied to the Thoracic Spine Improve Oxygen Saturation Levels and Thoracic Kyphosis in E-Cigarette Smokers?
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYIT-IRB-2025-299
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Kyphosis
Keywords: Thoracic spine, pulse oximetery, mobilzation

STUDY DESIGN:
Intervention Model Description: Experimental group will serve as their own control after a one-week washout period.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will not have knowledge of each participant's intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thoracic Mobilization (Experimental): The intervention group will receive a posterior to anterior directed thoracic mobilization to the mid-thoracic spine to facilitate extension. This will be imparted for a duration of 60 seconds, and this will be repeated for a total of three times. Interventions will be performed in a seated position.
  Interventions: Other: Thoracic Mobilization
- Light Touch Contact (Sham Comparator): The sham treatment will be applied to each subject. The sham treatment of light, non-therapeutic touch will be applied to both scapulae for three minutes. Interventions will be performed in a seated position.
  Interventions: Other: Light Touch Contact

INTERVENTIONS:
Other: Thoracic Mobilization — The intervention group will receive a posterior to anterior directed thoracic mobilization to the mid-thoracic spine to facilitate extension. This will be imparted for a duration of 60 seconds, and this will be repeated for a total of three times. Interventions will be performed in a seated position.
  Arms: Thoracic Mobilization
Other: Light Touch Contact — The sham treatment will be applied to each subject. The sham treatment of light, non-therapeutic touch will be applied to both scapulae for three minutes. Interventions will be performed in a seated position.
  Arms: Light Touch Contact

SUMMARY:
The goal of this study is to determine if manual therapy can improve thoracic spinal posture and pulse oximetery in individuals who use e-cigarettes.

The main questions the study aims to answer are:

* Is there an immediate improvements in thoracic posture
* Is there immediate improvements in pulse oximetery Research will compare an experimental group and a control group to examine the effects.

DETAILED DESCRIPTION:
All participants will be recruited from flyers posted throughout the NYIT Long Island campus. The participants will be screened for inclusion using set criteria by the PI.

In this crossover design study, participants will be randomly assigned to either an intervention experimental group or sham control group. The intervention group will received a thoracic extension mobilization to the mid-thoracic spine for a duration of 60 seconds and this will be repeated for a total of three times. The sham group will received a light, non-therapeutic touch to both scapulae which will be applied for three minutes. Both interventions will be performed in a seated position. Measurements of thoracic kyphosis and oxygen saturation will be taken before and after each procedure using inclinometers and a pulse oximeter, respectively.

After a washout period of one week, the participants will be return and receive the other form of intervention that they did no receive in in the first week. All procedures and outcomes will be performed as noted above.

ELIGIBILITY:
Inclusion Criteria:

Current e-cigarette user Accentuated thoracic kyphosis (Cobb angle >20 degrees) Age range: at least 18 years old Good overall health

Exclusion Criteria:

History of respiratory disease Recent vertebral fractures Recent spinal surgery Vertebral instability Congenital or acquired thoracic cage deformities Prolonged steroid use Osteoporosis/osteoporosis Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Angle of Thoracic Kyphosis | Immediately before and after each intervention
  Measurement of the thoracic kyphosis will be made both pre and post treatment using excepted normative values (Cobb angle)

SECONDARY OUTCOMES:
Oxygen Saturation | immediately before and after intervention
  Percentage of oxygen found in the peripheral circulation using a pulse oximeter

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M Ingenito, DPT, Principal Investigator — New York Institute of Technology
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD for this study.